CLINICAL TRIAL: NCT03630289
Title: Tissue Autograft to Bypass the Blood Brain Barrier (BBB) in Human Glioblastoma Multiforme (GBM)
Brief Title: Surgical Tissue Flap to Bypass the Blood Brain Barrier in GBM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, John Boockvar, MD Zucker SOM @Hofstra/Northwell, Principal Investigator, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-0498
Record Dates: First submitted 2018-08-02; First posted 2018-08-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Glioblastoma; Glioblastoma Multiforme; GBM; Brain Cancer
Keywords: tissue autograft; blood brain barrier
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical tissue autograft: TPF flap/pericranial flap (Experimental): Use of a pedicled autologous piece of tissue called the temporoparietal fascial (TPF) flap or pericranial flap into the resection cavity of newly diagnosed glioblastoma multiforme (GBM) patients
  Interventions: Procedure: Tissue autograft of pedicled temporoparietal fascial (TPF) or pericranial flap to bypass the blood brain barrier (BBB)

INTERVENTIONS:
Procedure: Tissue autograft of pedicled temporoparietal fascial (TPF) or pericranial flap to bypass the blood brain barrier (BBB) — Surgical tissue autograft of pedicled temporoparietal fascial (TPF) or pericranial flap into the resection cavity of newly diagnosed glioblastoma multiforme (GBM) patients.
  Other Names: surgical tissue flap; tissue autograft

SUMMARY:
This study assesses the safety of using tissue autograft of a pedicled temporoparietal fascial (TPF) or pericranial flap into the resection cavity of newly diagnosed glioblastoma multiforme (GBM) patients.

The objective of the study is to demonstrate that this surgical technique is safe in a small human cohort of patients with resected newly diagnosed GBM and may improve progression-free survival (PFS).

DETAILED DESCRIPTION:
Glioblastoma (GBM) is the most common primary central nervous system malignancy in adults, and accounts for over half of all malignant brain tumors. The prognosis for newly diagnosed GBM is extremely poor even with Stupp protocol consisting of surgery followed by temozolomide and radiotherapy. Present therapies are inadequate, as evidenced by the low 5-year survival rate for brain cancer patients, with median survival at approximately 12 months and treatment for GBM remains a significant unmet clinical need in oncology.

All subjects included in the study will initially undergo standard surgical resection for newly diagnosed GBM. Following the resection, the surgical cavity will be lined with a long pedicled, autologous piece of tissue called a temporoparietal fascial flap or pericranium. The patient's dura, bone and scalp will be closed as is customary. The permeability of the blood vessels of the TPF or pericranial flap should allow for improved delivery of therapeutics and immune cells (macrophages and T cells) into the vicinity, extracellular space and microenvironment of the resected tumor cavity including the brain adjacent to the GBM. The TPF or pericranial flap would easily conform to many resected GBM cavities in our human patients with acceptable risk. The TPF and pericranial flap with its predictable and rich vascular anatomy have been shown to be an ideal flap for cases of previously irradiated and/or infected wound beds.

The investigators hypothesize that a TPF or pericranial flap that is harvested in our patients with resected GBM may be used as a readily available and accessible means of circumventing the blood brain barrier selectively and focally. The investigators aim to prove that this surgical technique is safe in a small human cohort of patients with resected newly diagnosed GBM and may improve progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or female 18 years of age or older.
* Subject is undergoing planned resection of known or suspected GBM.
* Subject has a Karnofsky Performance Status (KPS) 70% or greater.
* Subject has a life expectancy of at least 6 months, in the opinion of the Investigator.
* Based on the pre-operative evaluation by neurosurgeon, the subject is a candidate for ≥ 80% resection of enhancing region.
* Subject must be able to undergo MRI evaluation.
* Subject meets the following laboratory criteria:

  * White blood count ≥ 3,000/µL
  * Absolute neutrophil count ≥ 1,500/µL
  * Platelets ≥ 100,000/µL
  * Hemoglobin > 10.0 g/dL (transfusion and/or ESA allowed)
  * Total bilirubin and alkaline phosphatase ≤ 2x institutional upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x ULN
  * Blood urea nitrogen (BUN) and creatinine < 1.5 x ULN
* Females of reproductive potential must have a negative serum pregnancy test and be willing to use an acceptable method of birth control.
* Males of reproductive potential must be willing to use an acceptable method of birth control to ensure effective contraception with partner.
* Able to understand and willing to sign an institutional review board (IRB)-approved written informed consent document (legally authorized representative permitted).

Inclusion criteria considered during surgery:

* Subject has a histologically confirmed (frozen section) diagnosis of WHO Grade IV glioblastoma multiforme (GBM).
* TPFF and/or pericranial flap is technically feasible.

Exclusion Criteria:

* Subject, if female, is pregnant or is breast feeding.
* Subject has initiated chemotherapy or radiation treatment for diagnosis of or GBM.
* Subject intends to participate in another clinical trial.
* Subject intends to undergo treatment with the Gliadel® wafer at the time of this surgery.
* Subject has an active infection requiring treatment.
* Subject has radiographic evidence of multi-focal disease or leptomeningeal dissemination.
* Subject has a history of other malignancy, unless the patient has been disease-free for at least 5 years. Adequately treated basal cell carcinoma or squamous cell skin cancer is acceptable regardless of time, as well as localized prostate carcinoma or cervical carcinoma in situ after curative treatment.
* Subject has a known positive test for human immunodeficiency virus infection, or active hepatitis B or hepatitis C infection.
* Subject has a history or evidence of any other clinically significant disorder, condition or disease that would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety parameter: proportion of patients experiencing rapidly progressive disease as indicated by MRI using RANO Criteria | Study Day 1-180
  Increase in tumor size relative to baseline will be measured using RANO and assessed by MRI throughout study at 24 hours, 7 days, 30 days, 60 days, 90 days, 180 days. Rapidly progressive disease is defined as 25% growth relative to baseline.
Safety parameter: proportion of patients experiencing increase in seizures, stroke, and infection | Study Day 1-180
  Increase in seizures (defined as 15% relative to baseline), occurrence of a stroke, or occurrence of a severe infection will be determined throughout study at 24 hours, 7 days, 30 days, 60 days, 90 days, 180 days.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 6 months
  The proportion of patients who are alive at 6 months from flap implantation and are progression-free will be estimated using standard methods for proportions, along with the associated exact 95% confidence interval. All patients will be followed for a minimum of six months from the time of implantation. For this analysis, patients who are lost to follow-up prior to 6 months will be (conservatively) assumed as treatment failures at 6 months. The investigators will also estimate PFS using the Kaplan-Meier Product Limit Method. For this analysis, subjects who are alive and have not progressed as of the date of last follow-up will be considered censored.
Overall Survival (OS) | 2 years
  OS will be calculated as the time from treatment initiation (TPF implantation) to the time of death. Subjects who are alive as of the date of last follow-up will be considered censored for survival. OS will be analyzed using the Kaplan-Meier Product Limit Method.

CONTACTS AND LOCATIONS:
Overall Officials: John Boockvar, MD, Principal Investigator — Northwell Health
Locations (1):
- Lenox Hill Brain Tumor Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Doron O, Wong T, Ablyazova F, Singha S, Cavallaro J, Ben-Shalom N, D'Amico RS, Harshan M, McKeown A, Zlochower A, Langer DJ, Boockvar JA. Results from a first-in-human phase I safety trial to evaluate the use of a vascularized pericranial/temporoparietal fascial flap to line the resection cavity following resection of newly diagnosed glioblastoma. J Neurooncol. 2024 Jun;168(2):225-235. doi: 10.1007/s11060-024-04647-w. Epub 2024 Apr 26. PMID 38664311